CLINICAL TRIAL: NCT01563211
Title: Predictive Modelling of Short Term Outcomes Following Systemic Neo-adjuvant and Adjuvant Therapy in Breast Cancer Patients
Brief Title: Predictive Model of Therapy Outcomes in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 72393/271478/14/611; 11-LO-1644 (Other: London Chelsea Research Ethics Committee)
Record Dates: First submitted 2012-01-25; First posted 2012-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Toxicity From Medication (Endocrine Treatment and Chemotherapy) Given for Breast Cancer Treatment.
Keywords: breast cancer therapy; toxicity; side effect profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma/serum urine buffy coat - for purposes of DNA extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients receiving endocrine treatment for breast cancer: Patients who are treated with tamoxifen, anastrozole or letrozole before or after surgery for breast cancer.
- Patients receiving chemotherapy for breast cancer: Patients receiving FEC (5-FU, cyclophosphamide, epiribicin) or FEC-D (FEC for 3 cycles, followed by 3 cycles of docetaxel).

SUMMARY:
Patients with breast cancer, who are treated with curative intent, have a combination of surgery (excision of the tumor) and a course of medical therapy (chemotherapy or endocrine treatment). Both treatments are associated with significant side effects. Chemotherapy is associated with nausea, vomiting, hair loss and bone marrow suppression, whereas endocrine therapy is associated with arthritis and menopausal symptoms. Patients taking either chemotherapy or endocrine treatment may experience a range of side effects. The range and severity of side effects experienced vary from patient to patient. Little or nothing is known about the reason for this difference.

The aim of the investigators proposal is to develop a pretreatment test to identify patients who are likely to undergo moderate to severe side effects, and therefore help doctors and patients plan and optimize medical therapy. The pretreatment test will be based on identifying a metabolic profile which can differentiate those patients who are likely to have severe or moderate side effects from those with either no or mild side effects. To do this, the investigators will take urine and blood samples from patients before and after the administration of endocrine treatment or chemotherapy and generate metabolic profiles.

Furthermore, the investigators aim to gain an understanding into why side effects experienced between different patients are so variable. To do this the investigators plan to perform cytokine analysis, targeted genetic analysis and pharmaokinetic analysis on blood sample collected from patients before and after treatment has commenced. Patients who have planned surgical excision of tumor and are recommended to receive medical therapy before or after surgery would be invited to join the study. Each patient will be required to make additional visits to the hospital to complete questionnaires regarding side effects experienced and for sample (urine and blood) collection. The investigators plan to recruit 168 patients.

DETAILED DESCRIPTION:
Patients with breast cancer are treated with a combination of surgery and medical treatment (either before (neoadjuvant) or after (adjuvant) surgery). Eligible patients will be identified by the oncologist and from the multidisciplinary meeting.

Once eligible patients have been identified they will be informed of the study by their oncologist, and then approached by the research team who will give them a patient information leaflet, discuss the study, answer any questions and ask the patient to sign a consent form if they are would like to participate in the study. The consent form must be signed before any study related procedures are performed.

Patients who have had surgery prior to receiving medical treatment (i.e. patients planned to receive adjuvant treatment, or patients who have a sentinel lymph node biopsy prior to starting neoadjuvant treatment) will have blood and urine samples taken before they have their surgery, at the preassessment surgical appointment.

The week before the patient starts medical therapy (either chemotherapy or endocrine treatment) the patient will need to attend Charing Cross Hospital for the following procedures (this may be an extra visit, depending on hospital appointments):

* To see the study doctor for a medical history and physical examination
* Pulse and blood pressure measurements
* BMI (body mass index) and body fat assessment
* To fill out a quality of life (QOL) questionnaire with research staff
* Routine blood tests (for haematology and biochemistry)
* Blood sample for metabolic profiling and cytokine analysis
* Urine sample for metabolic profiling
* The blood taken will additionally be tested for targeted genetic analysis if the patient has consented for this (as this is optional)

The patient will be asked to return to Charing Cross Hospital 24 hours later after an overnight fast for (this will be an extra visit): • Fasted blood and urine samples for metabolic profiling.

It is important to get fasted samples from patients, as diet influences the metabolic profile. Therefore to try to eliminate diet as a confounder it is important to get a fasted sample. Additionally, at the time of collection of blood and urine samples for metabolic profile analysis patients will be asked when they last ate, what they last ate and any specific dietary preferences/requirements (i.e. vegetarian, gluten free diet).

Further tests differ depending on whether the patient is receiving chemotherapy or endocrine treatment.

Patients receiving chemotherapy have 6 cycles, each cycle last 21 days. There are two types of chemotherapy given for breast cancer which are FEC (6 cycles of 5fluorouracil, epirubicin and cyclophosphamide) or FECD (3 cycles of 5fluorouracil, epirubicin and cyclophosphamide followed by 3 cycles of docetaxel). Patients receiving all types of chemotherapy (FEC and FECD) patients will be required to attend at the following time for procedures are explained below:

* Cycle 1, day 2

  o 24 hours after the patient received their chemotherapy treatment we will take urine and blood samples for metabolic profiling, and blood samples for routine blood tests (haematology and biochemistry) and cytokine analysis.
  * At this time the patient will also be asked to fill out 2 questionnaires with research staff - the first will be adverse effects experienced (questions from CTCAEv4.0), and the second will be a QOL questionnaire.
  * This will be an extra visit.
* Cycle 2, day 1

  * Prior to receiving their next cycle of chemotherapy urine and blood samples will be taken for metabolic profiling. Blood samples will be taken for routine tests (haematology and biochemistry) and for cytokine analysis.
  * Two questionnaires (questionnaire based on adverse effects experienced and QOL questionnaire) will be completed with research staff.
  * A blood sample will be taken after 10 minutes chemotherapy infusion has finished. Pharmacokinetic analysis for 5FU will be conducted on this sample. If possible the sample will be taken from the cannula through which the chemotherapy medication was administered (the first 10mls will need to be discarded to avoid contamination).
  * This will not be an extra visit if there has been no change to planned This will not be an extra visit if there has been no change to planned treatment schedule. If patients have consented for optional pharmacokinetic analysis the following sample will also be taken.
* Cycle 2, day 1 (optional assessment)

  o Three blood samples will be taken during the following 4 hours for pharmacokinetic analysis of cylophosphamide and epirubicin. If possible all samples will be taken from the cannula through which the chemotherapy was administered.
* Cycle 2, day 2 (optional assessment) o A blood sample will be taken 24 hours after the chemotherapy was given for pharmacokinetic analysis of cyclophosphamide.
* Cycle 2, day 3 (optional assessment)

  o A blood sample will be taken 48 hours after the chemotherapy was given for pharmacokinetic analysis of epirubicin.
* Cycle 6, day 21

  * Two questionnaires (questionnaire based on adverse effects experienced and QOL questionnaire) will be completed with research staff.
  * BMI (body mass index) and body fat assessment.
  * This will be an extra visit.

If patients are on FECD chemotherapy, they will attend at the above time points, but they will additionally be asked to attend after their docetaxel has commenced. This is required to test whether docetaxel has a different reaction in the body to the previous chemotherapy given. Patients will be asked to attend at the following time points for the following procedures:

* Cycle 4, day 2

  o 24 hours after the patient received their chemotherapy treatment we will take urine and blood samples for metabolic profiling, and blood samples for routine blood tests (haematology and biochemistry) and cytokine analysis.

  o Two questionnaires (questionnaire based on adverse effects experienced and QOL questionnaire) will be completed with research staff

  o This will be an extra visit
* Cycle 5, day 1

  * Prior to receiving their next cycle of chemotherapy urine and blood samples will be taken for metabolic profiling. Blood samples will be taken for routine tests (haematology and biochemistry) and for cytokine analysis.
  * Two questionnaires (questionnaire based on adverse effects experienced and QOL questionnaire) will be completed with research staff.
  * This will not be an extra visit if there has been no change to planned treatment schedule.

If patients have consented for optional pharmacokinetic analysis the following sample will also be taken.

• Cycle 5, day 1

o A blood sample will be taken at the end of the chemotherapy infusion and 6 hours after the infusion completed. If possible the blood samples will be taken from the cannula (the first 10mls taken from the cannula will need to be discarded to avoid contamination).

Patients receiving endocrine treatment will be asked to attend at the following time points after starting treatment for procedures listed below, in addition to baseline assessments described above:

* Day 2

  * Urine and blood samples for metabolic profiling. Blood samples for routine tests (haematology and biochemistry) and cytokine analysis.
  * This will be an extra visit
* Day 21

  * Two questionnaires (questionnaire based on adverse effects experienced and QOL questionnaire) will be completed with research staff.
  * Urine and blood samples for metabolic profiling. Blood samples for routine tests (haematology and biochemistry) and cytokine analysis.
  * This will be an extra visit
* At 5 months

  * Two questionnaires (questionnaire based on adverse effects experienced and QOL questionnaire) will be completed with research staff.
  * BMI (body mass index) and body fat assessment.
  * A blood sample for pharmacokinetic analysis
  * This will be an extra visit

All procedures and interviews will be conducted at Charing Cross Hospital. All patients will be enrolled in the study for 5 months. However, for patients receiving chemotherapy, if there has been a change in treatment schedule by the oncologist the time the patient will spend in the study will be increased in accordance with changes made to treatment schedule (i.e. if cycle 4 (docetaxel) is started 1 week late, then the time in the study will be 5 months and 1 week).

For patients receiving neoadjuvant treatment (chemotherapy or endocrine treatment before surgery) we will look at imaging and pathology reports to establish how the tumour has responded to treatment.

We aim to recruit 168 patients, 84 receiving endocrine therapy (either an oestrogen receptor antagonist or aromatase inhibitor) and 84 receiving cytotoxic chemotherapy (FEC or FECD).

The study will be conducted in 5 phases:

1. Patient recruitment and collection of samples (months 112)
2. H NMR spectroscopic analysis and UPLMS analysis of samples (months 718)
3. Mathematical modelling of the data (months 120)
4. Structural identification of candidate biomarkers (months 1822)
5. Write up of results and guidelines (months 2024)

The results will be analysed and published (in both presentations and a peer reviewed journal) at the end of the study. No patient identifiable information will be present in these publications. As all tests are carried out for research purposes and will be of no direct benefit to patients participating in this study, there are no plans to inform patients of their individual results. Patients will be informed of the overall results from the study that may result in a publication.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven breast cancer.
* Female ≥ 18 years of age, no upper age limit.
* Pretreatment haematology and biochemistry values with acceptable limits:
* Haemoglobin (Hb) > 9g/dl
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤ 1.5 x ULN
* Serum bilirrubin ≤ 1.5 x ULN
* Alkaline phosphatase ≤ 1.5 x ULN
* White blood cell (WBC) count ≥ 3.0 x 109/L and absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Serum creatinine ≤ 1.5 x ULN
* WHO performance status 0 or 1
* No active or uncontrolled infection
* Written informed consent prior to commencement of specific protocol procedures
* No concomitant medical, psychiatric or geographical problems that might prevent follow up of symptoms according to protocol.

Exclusion Criteria:

* Other serious illness or medical condition:
* Congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year prior to study entry, uncontrolled hypertension or high risk of uncontrolled arrhythmias
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizure that would prohibit the understanding and giving of informed consent
* Active uncontrolled infection
* Active peptic ulcer, unstable diabetes mellitus
* Only cytological proof of malignancy
* Patients not able or willing to give informed consent
* Patients taking medication other than low dose aspirin, antihypertensives or statins.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have newly diagnosed primary breast cancer who will be receiving chemotherapy (FEC and FEC-D regimes only) or endocrine treatment (anastrozole, letrozole or tamoxifen only).
  All new patients with Breast Cancer are discussed at the multidisciplinary team meeting (MDT) where they will be identified for the study. Patients will be identified by the oncologist and the multidisciplinary team (i.e the existing clinical care team).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for the study is to determine the relationship between metabonomics spectrum and side effects from chemotherapy and endocrine therapy for patients receiving treatment for breast cancer. | 2 years
  To identify a pre-treatment metabolic profile to predict patients who will experience moderate to severe side effects.

SECONDARY OUTCOMES:
Conduct pharmokinetic analysis of drugs administered and determine relationship between pharmacokinetics and severity of side effects experienced. | 2 years
  Measure pharmokinetics of each drug to try and ascertain underlying reasons for differences in toxicity.
Conduct cytokine analysis pre and post treatment, to determine relationship with severity of side effects experienced. | 2 years
Conduct targeted genetic analysis to determine relationship with severity of side effects experienced. | 2 years
  To identify known SNPs implicated in toxicity to metabolic profile/biomarkers found.
To find underlying mechanism to explain the interpatient variability in severity of side effects experienced using above techniques (i.e. metabolic profile, pharmacokinetic analysis, cytokine analysis and targeted genetic analysis). | 2 years
To identify a biomarker based on metabnomic profiling for response to treatment for those receiving neoadjuvant treatment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Coombes, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom